CLINICAL TRIAL: NCT02959164
Title: A Phase 1b Study: Treatment of Refractory Pancreatic Adenocarcinoma and Advanced Soft Tissue or Bone Sarcomas Using Decitabine Combined With Gemcitabine
Brief Title: Decitabine and Gemcitabine for Pancreatic Cancer and Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201610750
Record Dates: First submitted 2016-11-06; First posted 2016-11-08 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Decitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine and Gemcitabine (Experimental): Decitabine, Dose escalation starting at 0.1mg/kg, subcutaneously administered on twice weekly schedule for three weeks of a 28 day cycle.
  Gemcitabine fixed infusion rate of 900 mg/m2, IV over 90 min, on Days, 1, 8 and 15 of a 28-day cycle.
  Interventions: Drug: Decitabine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Decitabine — Dose escalation starting at 0.1mg/kg, subcutaneously administered on twice weekly schedule for three weeks of a 28 day cycle.
  Dose Escalation Schedule Dose Level/Dose of Decitabine per cycle Level -2: 0.1 mg/kg SQ twice weekly for 1 week; Level -1: 0.1 mg/kg SQ twice weekly for 2 weeks; Level 1*: 0.1 mg/kg SQ twice weekly for 3 weeks; Level 2: 0.2 mg/kg SQ twice weekly for 3 weeks;
  *Starting Dose Level
  Other Names: Dacogen
Drug: Gemcitabine — Fixed infusion rate of 900 mg/m2, IV over 90 min, on Days, 1, 8 and 15 of a 28-day cycle.
  Dose Escalation Schedule Dose Level/Dose of Decitabine per cycle Level -2: 0.1 mg/kg SQ twice weekly for 1 week; Level -1: 0.1 mg/kg SQ twice weekly for 2 weeks; Level 1*: 0.1 mg/kg SQ twice weekly for 3 weeks; Level 2: 0.2 mg/kg SQ twice weekly for 3 weeks;
  *Starting Dose Level
  Other Names: Gemzar

SUMMARY:
The purpose of this Phase 1b study is to assess the safety and maximum tolerated dose (MTD) of Decitabine in combination with Gemcitabine among previously treated patients diagnosed with advanced pancreatic adenocarcinoma or sarcoma (soft tissue and bone).

DETAILED DESCRIPTION:
The objectives of this study are to assess the safety and tolerability of the combination of Decitabine with Gemcitabine in previously treated patients with advanced pancreatic cancer and advanced sarcoma and to define the recommended Phase II dose and describe the dose-limiting toxicity of the combination of Decitabine with Gemcitabine. The preliminary efficacy parameters of the combination of Decitabine with Gemcitabine will be estimated in terms of response rate, disease control rate and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have metastatic histologically or cytologically confirmed pancreatic adenocarcinoma or sarcoma (soft tissue or bone). Patient may enroll if he or she refuses first line therapy.
2. Age ≥18 years.
3. ECOG performance status ≤2 (Karnofsky ≥60% (See Appendix 1).
4. Life expectancy of greater than 3 months (does not apply to pancreatic cancer population).
5. Measureable disease per RECIST criteria.
6. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count ≥1,500/mm3
   * Platelets ≥100 k/mm3
   * Total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
   * Creatinine </= 1.5 ULN
7. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) from time of consent and for the duration of study participation as well as for 3 months after the completion of study drug. Adequate contraception consists of a double method of contraception, one method of which must be a barrier method.

   WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).

   If a woman (or a male subject's female partner) becomes pregnant or suspects she is pregnant while she is participating in this study, she should inform her treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Chemotherapy or radiotherapy within 4 weeks (for targeted therapies 5 half-lives) prior to entering the study or failure to recover from adverse events due to agents administered to </= grade 1 or stable grade 2, at the discretion of the treating physician.
2. Patients who are receiving any other investigational agents.
3. Known brain metastases.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Decitabine or other agents used in study.
5. Prior Decitabine for the treatment of this cancer. Patients with previous exposure to therapy with Gemcitabine are allowed in the study.
6. Pregnant or breast feeding women are excluded from participating in this study. WOCBP must have a negative serum pregnancy test within 7 days of the first administration of Decitabine.
7. Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required.
8. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity - To examine the toxicity related to the therapy by measuring the number of treatment related adverse events in patients | All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s) up to 30 days after the last date of any study therapy
  Non-Hematologic - Any grade 3,4 solid organ toxicity not explainable by another cause in the opinion of the principal investigator
Tumor Response Rate - Change at evaluations | Change on two consecutive evaluations at least 8 weeks apart up to 30 days after the last date of any study therapy
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Patients will be evaluated weekly during each cycle of treatment up to 30 days after the last date of any study therapy
  DCR is defined as the proportion of patients who achieved a complete response (CR), partial response (PR) or stable disease (SD).
Progression-free survival (PFS) | Patients will be evaluated weekly during each cycle of treatment up to 30 days after the last date of any study therapy
  PFS is defined as the duration of time from start of treatment to time of progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Patients will be evaluated weekly during each cycle of treatment up to 30 days after the last date of any study therapy
  OS is defined as the duration of time from start of treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02959164/ICF_000.pdf